CLINICAL TRIAL: NCT03557684
Title: An Experimental Treatment Approach for Inflammation-Induced Depression
Brief Title: Leucine for Depression Study (L-DEP)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Hyong-Jin Cho, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R21MH113915 (NIH); R21MH113915 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Leucine; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PO leucine & IV LPS (Experimental): Oral (PO) leucine 6 g twice a day for 2 weeks followed by a single intravenous (IV) bolus of lipopolysaccharide (LPS) 0.8 ng/kg of body weight
  Interventions: Dietary Supplement: leucine; Biological: lipopolysaccharide (LPS)
- PO placebo & IV LPS (Experimental): PO maltodextrin (placebo) twice a day for 2 weeks followed by a single IV bolus of LPS 0.8 ng/kg of body weight
  Interventions: Other: PO placebo; Biological: lipopolysaccharide (LPS)
- PO leucine & IV placebo (Experimental): PO leucine 6 g twice a day for 2 weeks followed by a single IV bolus of 0.9% saline
  Interventions: Dietary Supplement: leucine; Other: IV placebo
- PO placebo & IV placebo (Placebo Comparator): PO maltodextrin (placebo) twice a day for 2 weeks followed by a single IV bolus of 0.9% saline
  Interventions: Other: PO placebo; Other: IV placebo

INTERVENTIONS:
Dietary Supplement: leucine — amino acid leucine in powder
  Arms: PO leucine & IV LPS; PO leucine & IV placebo
Other: PO placebo — maltodextrin
  Arms: PO placebo & IV LPS; PO placebo & IV placebo
Biological: lipopolysaccharide (LPS) — purified bacterial wall component as an inflammatory challenge
  Arms: PO leucine & IV LPS; PO placebo & IV LPS
Other: IV placebo — 0.9% saline
  Arms: PO leucine & IV placebo; PO placebo & IV placebo

SUMMARY:
Depression is very common and poses a huge disease burden. About 20% of the US population suffers from depression at lease once in their lifetime. Inflammations that are hidden inside our body as a result of aging, obesity, chronic diseases, or certain treatments (e.g., interferon for hepatitis C) appear to cause depressive symptoms and even clinical depression. Individuals with such inflammations are more likely to suffer from depression and are less likely to respond to currently available antidepressant medications. This study will test leucine, an amino acid, as a new way to mitigate depressive symptoms in response to such inflammations. This study begins with a 90-minute screening session to determine whether participants are eligible to join the main study. Those who meet the eligibility criteria will then join the main study, which will consist of taking leucine or maltodextrin (i.e., oral placebo) for 2 weeks at home and an 8-hour session at the UCLA Medical Center. A brief telephone follow-up every 3 months for 2 years with questions on mood is also planned. Approximately 90 healthy adults will be recruited for participation in the study. During the course of the study, participants will take leucine or maltodextrin for 2 weeks at home and then will be injected either lipopolysaccharide (LPS) or saline (i.e., intravenous placebo) at the UCLA Medical Center. LPS is a bacterial substance that can initiate chemical reactions that are similar to those seen in individuals with mild sickness symptoms, such as a slight increase in body temperature, muscle aches, or tiredness. It is a safe way of investigating the body's response to inflammation and how these changes may alter cognitive, emotional, or neural function. It has been given thousands of times to healthy volunteers - both younger and older adults - without any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

Participants will be required to be in good general health (as evaluated during the phone and in-person screening sessions) and aged 18 to 65 years.

Exclusion Criteria:

Following a structured telephone interview, prospective participants with the following conditions will not advance to the in-person screening session: presence of chronic mental or physical illness, history of allergies, autoimmune, liver, or other severe chronic diseases, current use of prescription medications such as steroids, NSAIDs, immune modifying drugs, opioid analgesics, and psychotropics, or previous history of fainting during blood draws. These inclusion and exclusion criteria will be examined in detail and confirmed in the in-person screening session by the study physician. Furthermore, any participant who has any of the following conditions will be ineligible for the study. Medical Conditions: (1) presence of co-morbid medical conditions not limited to but including maple syrup urine disease (a contraindication to leucine treatment), cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders; (2) presence of co-morbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders; (3) presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk; (4) presence of chronic infection, which may elevate proinflammatory cytokines; (5) presence of an acute infectious illness in the two weeks prior to the screening session. Psychiatric Disorders: (6) an Axis I psychiatric disorder as determined by the Research Version of the Structured Clinical Interview for DSM-5 (SCID-5-RV) including a current major depressive disorder (a prior history of depression is not an exclusion criterion, which will be considered for a pre-planned sensitivity analysis); (7) lifetime history of suicide attempt or inpatient psychiatric admission; (8) current suicidal ideation assessed by the Columbia Suicide Severity Rating Scale (C-SSRS); (9) current depressive symptoms assessed by the PHQ-9 (≥ 5)). Medication and Substance Use: (10) current and/or past regular use of hormone-containing medications including steroids; (11) current and/or past regular use of non-steroid anti-inflammatory drugs; (12) current and/or past regular use of immune modifying drugs that target specific immune responses such as TNF antagonists; (13) current and/or past regular use of analgesics such as opioids; (14) current and/or past regular use of psychotropic medications, including antidepressants, anxiolytics, antipsychotics, hypnotics, sedatives, and barbiturates; (15) current and/or past regular use of cardiovascular medications, including antihypertensive, antiarrhythmic, antianginal, and anticoagulant drugs; (16) current smoking or excessive caffeine use (>600 mg/day) because of the known effects on proinflammatory cytokine levels; (17) evidence of recreational drug use from urine test. Health Factors: (18) BMI > 35 because of the effects of obesity on proinflammatory cytokine activity and also on risk for sleep disordered breathing; or (19) any abnormalities on screening laboratory tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua H Cho, MD, PhD, Principal Investigator — University of California Los Angeles David Geffen School of Medicine
Locations (1):
- UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 88 subjects were interviewed, 73 eligible, and 70 randomized. Out of these 70, 11 did not participate in the actual study (7 declined; 3 tested positive in urine toxicology on the study day, which was a pre-set exclusion criterion; 1 reported using a drug given by another study on the study day). Thus, 59 were enrolled in and started the study, an experimental provocation trial involving LPS injection, which was a necessary step for a participant to be considered enrolled and started.
Period: Overall Study
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Started | 23 | 18 | 8 | 10
Completed | 23 | 18 | 8 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo | Total
Number analyzed (Participants) | 23 | 18 | 8 | 10 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (16.3) | 26.8 (12.7) | 33.1 (12.6) | 31.9 (14.9) | 31.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 2 | 4 | 24
  Male | 13 | 10 | 6 | 6 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 1 | 8
  Not Hispanic or Latino | 19 | 17 | 6 | 9 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 9 | 1 | 3 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 10 | 8 | 6 | 7 | 31
  More than one race | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 18 | 8 | 10 | 59
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.3 (4.0) | 23.6 (3.0) | 26.3 (2.9) | 25.5 (4.0) | 24.6 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressed Mood From Baseline
Description: Depression Subscale of the Short Form of the Profile of Mood States (POMS-SF): total score ranges from 0 to 32; higher values represent worse outcome, i.e., more severe depressed mood; the absolute values at each time point are presented here rather than change of values between time points; zero (0) in mean and standard deviation reflect measured data and not placeholder values.
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Baseline | .6818182 (1.86155) | .5294118 (1.178858) | .2857143 (.48795) | .6 (1.074968)
  1 hour | 1.619048 (3.879126) | .7647059 (1.480262) | .375 (.7440238) | 0 (0)
  1.5 hours | 1.55 (3.817894) | 1 (2.371708) | .25 (.46291) | .1 (.3162278)
  2 hours | 1 (3.829708) | 1.111111 (3.103866) | .7142857 (1.253566) | .4 (.6992059)
  3 hours | .5909091 (2.363595) | .5625 (1.364734) | .375 (1.06066) | .1111111 (.3333333)
  4 hours | .4285714 (1.963961) | .3333333 (.9701425) | .1428571 (.3779645) | 0 (0)
  5 hours | .4545455 (2.132007) | .0555556 (.2357023) | .1666667 (.4082483) | 0 (0)
  6 hours | .5238095 (2.182179) | 0 (0) | .1428571 (.3779645) | 0 (0)

2. Secondary Outcome: Change in Depressive Symptoms From Baseline
Description: Montgomery-Asberg Depression Rating Scale (MADRS): a clinician-rated questionnaire of depressive symptoms with scores ranging from 0 to 60, with higher scores indicating more severe depressive symptoms.
Time Frame: At baseline and then at 2 and 4 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Baseline | 2.086957 (2.574579) | 2.125 (3.052322) | 2.5 (3.891382) | 1.222222 (1.301708)
  2 hours | 3 (5.485913) | 4 (6.184658) | 1.875 (2.295181) | .7 (.9486833)
  4 hours | 1.045455 (1.812057) | 1.529412 (1.907801) | 2.142857 (1.864454) | .2 (.421637)

3. Secondary Outcome: Change in Feelings of Social Disconnection From Baseline
Description: Feelings of Social Disconnection Scale: a self-report questionnaire of feelings of social disconnection with scores ranging from 0 to 28, with higher scores indicating more severe feelings of social disconnection.
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Baseline | 22.52381 (7.639496) | 24 (8.581786) | 22.57143 (6.704654) | 21.6 (10.7827)
  1 hour | 16.65217 (7.327462) | 17.83333 (9.463552) | 18 (6.21059) | 15.44444 (12.26898)
  1.5 hours | 16.86364 (7.942025) | 16.77778 (9.42809) | 17.125 (6.220645) | 13.625 (7.836499)
  2 hours | 15.33333 (7.308335) | 17.05556 (9.276613) | 17 (6.546537) | 18.3 (14.95215)
  3 hours | 15.38095 (6.6744) | 15.8125 (9.914426) | 18 (5.744563) | 13.55556 (9.166667)
  4 hours | 15.71429 (7.26046) | 16.66667 (9.749811) | 16.42857 (6.803361) | 19.6 (19.65932)
  5 hours | 16.28571 (7.444077) | 19.38889 (13.3775) | 19.5 (10.96814) | 17.6 (14.19859)
  6 hours | 16.25 (7.27559) | 17.72222 (8.68945) | 14.57143 (7.807201) | 19.9 (18.62167)

4. Secondary Outcome: Change in Fatigue From Baseline
Description: Fatigue Subscale of the Short Form of the Profile of Mood States (POMS-SF): total score ranges from 0 to 20; higher values represent worse outcome, i.e., more severe fatigue; the absolute values at each time point are presented here rather than change of values between time points.
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Baseline | 2.409091 (2.839502) | 2.117647 (2.027386) | 1.857143 (3.338092) | 2 (1.885618)
  1 hours | 3.666667 (4.09064) | 3.611111 (3.310214) | 2.25 (3.412163) | .6666667 (.8660254)
  1.5 hours | 5.095238 (5.290603) | 4.444444 (2.994548) | 2.25 (4.399675) | 1 (1.247219)
  2 hours | 4.681818 (5.083928) | 4.333333 (3.694193) | 2.375 (3.73927) | .9 (1.449138)
  3 hours | 4.590909 (4.584229) | 3.555556 (3.014128) | 2.625 (4.10357) | 1.777778 (1.855921)
  4 hours | 3.272727 (4.322497) | 2.111111 (2.246275) | 2.571429 (4.197505) | .6 (1.074968)
  5 hours | 3.454545 (4.925418) | 2.222222 (2.438793) | 2.833333 (4.167333) | 1.3 (1.946507)
  6 hours | 2.666667 (4.564355) | 1.944444 (2.508157) | 1.571429 (2.935821) | 1 (1.581139)

5. Secondary Outcome: Change in Confusion From Baseline
Description: Confusion Subscale of the Short Form of the Profile of Mood States (POMS-SF): total score ranges from 0 to 20; higher values represent worse outcome, i.e., more severe confusion; the absolute values at each time point are presented here rather than change of values between time points; zero (0) in mean and standard deviation reflect measured data and not placeholder values.
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Baseline | 1.409091 (1.991867) | 1.125 (1.408309) | 1 (1.825742) | 1.1 (1.286684)
  1 hours | 2.238095 (3.845839) | .8888889 (1.07861) | 1 (1.414214) | .4444444 (1.013794)
  1.5 hours | 2.095238 (3.462727) | 1.222222 (1.308594) | .375 (1.06066) | .1 (.3162278)
  2 hours | 1.772727 (3.435554) | 1.111111 (1.323493) | .625 (1.407886) | .1 (.3162278)
  3 hours | 1.454545 (2.063914) | .8888889 (1.131833) | .625 (1.06066) | .3333333 (.7071068)
  4 hours | .6363636 (1.216766) | .6111111 (1.195033) | .5714286 (1.133893) | 0 (0)
  5 hours | .6363636 (1.398824) | .6111111 (1.036901) | .5 (.5773503) | .1 (.3162278)
  6 hours | .4761905 (1.435933) | .4705882 (1.06757) | .1428571 (.3779645) | 0 (0)

6. Secondary Outcome: Change in Memory Domains of Cognitive Function From Baseline
Description: Memory domains of cognitive function were measured using the computerized tests from CNS Vital Signs™: verbal memory using "Verbal Memory Test" (total scores ranging from 0 to 60; higher scores mean a better outcome); and visual memory using "Visual Memory Test" (total scores ranging from 0 to 60; higher scores mean a better outcome). The absolute values at each time point are presented.
Time Frame: At baseline and then 3 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
score on a scale
  Verbal memory baseline | 51.30435 (8.298054) | 53.23529 (6.139314) | 51.125 (4.580627) | 52.3 (8.525126)
  Verbal memory 3 hours | 48.66667 (5.695027) | 52.58824 (6.538911) | 48.5 (5.976143) | 45.5 (10.31988)
  Visual memory baseline | 44.04348 (6.588408) | 47.76471 (5.695716) | 46.125 (6.490377) | 43.9 (8.736259)
  Visual memory 3 hours | 42.2381 (6.106593) | 46.29412 (7.405781) | 41.75 (4.26782) | 40.9 (9.097619)

7. Other Pre Specified Outcome: Anhedonia
Description: Facial expressions and skin conductance in response to funny film clips using the iMotions®Attention Tool (iMotions Inc., Cambridge, MA) which performs automatic analysis of facial expressions from video and integrates simultaneous measurement of skin conductance
Time Frame: 2 hours after LPS (or saline) administration
Population: The study was paused during the COVID pandemic because endotoxin, a biologic derived from an infectious agent, was being used. Then, the request for COIVD supplement to NIMH was denied, and due to the lack of funds, the study was prematurely terminated. As the raw data of this particular outcome measure consist in recordings of facial expression and skin conductance, further processing by a specialized technician and additional funds are required. Thus we are currently unable to report the data.
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Subjective Sensitivity to Social Rejection
Description: Using the Cyberball Social Exclusion Task, feelings of social distress to social rejection are evaluated based on a scale with the total score ranging from 0 to 48; higher values represent worse outcome, i.e., more severe social distress. The Overall Number of Participants Analyzed is different from numbers of participants reported in the Participant Flow module because some participants declined to complete this task.
Time Frame: 2 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 20 | 17 | 8 | 10
score on a scale | 18.05 (5.670561) | 16.17647 (5.282463) | 18.25 (7.245688) | 17.6 (5.481281)

9. Other Pre Specified Outcome: Negative Bias in Facial Emotion Recognition
Description: Emotional Face Recognition Task consists in showing participants a series of black and white photographs (Ekman Pictures of facial affect), in which the facial expression is morphed from neutral to either Sad, Angry, or Happy. For each image, participants will be asked to make a forced choice about the emotion expressed, and rate their certainty.
Time Frame: 2 hours after LPS (or saline) administration
Population: The study was paused during the COVID pandemic because endotoxin, a biologic derived from an infectious agent, was being used. Then, the request for COIVD supplement to NIMH was denied, and due to the lack of funds, the study was prematurely terminated. As the raw data of this particular outcome measure require further processing by a specialized technician and thus additional funds, we are currently unable to process and report the data.
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Subjective Sensitivity to Social Acceptance
Description: Prior to the experimental session, participants are asked to complete a survey that contains several personality questionnaires and are video-recorded for 2-5 minutes as they discuss what they like about themselves. Participants are told that 8 people will form impressions of them by selecting personality traits to describe them. Participants then see a photograph of themselves along with a descriptive word underneath (supposedly provided by the evaluators), which is pre-rated based on desirability, and are asked to rate subjective happiness when each of the feedback items is presented. The total score of the scale ranges from 0 to 105; higher values represent better outcome, i.e., higher social reward. The Overall Number of Participants Analyzed is different from numbers of participants reported in the Participant Flow module because some participants declined to complete this task.
Time Frame: 2 hours after drug administration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 21 | 18 | 7 | 10
score on a scale | 76.7619 (9.229869) | 77.38889 (5.94226) | 76.28571 (3.77334) | 78.3 (6.037844)

11. Other Pre Specified Outcome: Reward
Description: Reward Learning Task (a laboratory based probabilistic reward task that objectively measures participants' ability to modulate behavior as a function of reward)
Time Frame: 2 hours after LPS (or saline) administration
Population: as for outcome 9
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Change in Proinflammatory Cytokines From Baseline
Description: Plasma proinflammatory cytokines (interleukin-1 receptor antagonist, interleukin-6, tumor necrosis factor-α, and soluble tumor necrosis factor receptor)
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Population: The study was paused during the COVID pandemic because endotoxin, a biologic derived from an infectious agent, was being used. Then, the request for COIVD supplement to NIMH was denied, and due to the lack of funds, the study was prematurely terminated. As the raw data of this particular outcome measure require further processing and thus further funds, we are currently unable to process and report the data.
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Change in Kynurenine Metabolites From Baseline
Description: Plasma tryptophan, kynurenine, quinolinic acid, and kynurenic acid
Time Frame: At baseline and then at 1, 1.5, 2, 3, 4, 5, and 6 hours after LPS (or saline) administration
Population: The study was paused during the COVID pandemic because endotoxin, a biologic derived from an infectious agent, was being used. Then, the request for COIVD supplement to NIMH was denied, and due to the lack of funds, the study was prematurely terminated. Due to the lack of funds, the blood sample could not be assayed, and we are currently unable to report the data for this particular outcome measure.
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Change in Gene Expression From Baseline
Description: Genome-wide transcriptional profiling conducted using Illumina HT-12 BeadArrays
Time Frame: At baseline and 30 minutes after LPS (or saline) administration
Population: as for outcome 13
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Change in Non-memory Domains of Cognitive Function From Baseline
Description: Non-memory domains of cognitive function were measured using the computerized tests from CNS Vital Signs™: executive function using "Stroop Test" (average reaction time in milliseconds thus ranging from 0 to infinite; shorter reaction time means a better outcome); and attention using "Shifting Attention Test" (average reaction time for correct responses in milliseconds thus ranging from 0 to infinite; shorter reaction time means a better outcome) and "Continuous Performance Test" (average reaction time for correct responses in milliseconds thus ranging from 0 to infinite; shorter reaction time means a better outcome). The absolute values at each time point are presented.
Time Frame: At baseline and then 3 hours after LPS (or saline) administration
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
Number analyzed (Participants) | 23 | 18 | 8 | 10
milliseconds
  Stroop test baseline | 356.913 (95.80563) | 307.6471 (57.51515) | 304.125 (38.96679) | 268.8 (146.5619)
  Stroop test 3 hours | 386.2381 (93.90842) | 316.2353 (53.88475) | 324.25 (36.86946) | 337.4 (45.80442)
  Shifting attention baseline | 1014.174 (199.4204) | 899.6471 (140.7502) | 935.75 (185.7423) | 947.9 (140.4457)
  Shifting attention 3 hours | 957.2857 (211.8759) | 829.7647 (131.7823) | 943 (109.6696) | 957.5 (156.2358)
  Continuous performance baseline | 449.1304 (73.88954) | 426 (44.63743) | 442.25 (27.41089) | 458.2 (44.96122)
  Continuous performance 3 hours | 456.619 (65.31422) | 423.8235 (54.88993) | 439.25 (35.05812) | 460.6 (55.05795)

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | PO Leucine & IV LPS | PO Placebo & IV LPS | PO Leucine & IV Placebo | PO Placebo & IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/18 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/23 | 0/18 | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT03557684/Prot_SAP_000.pdf